CLINICAL TRIAL: NCT04444401
Title: InterNaTional rEgistry oN Sars-cov-2posItiVe nEuroendocrine Neoplasm Patients (INTENSIVE)
Brief Title: Registry on NEN Patients and COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: IEO-1291
Record Dates: First submitted 2020-06-22; First posted 2020-06-23 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Neuroendocrine Tumors; COVID-19
Keywords: NEN; NET; NEC; COVID-19; SARS-CoV-2; Coronavirus
MeSH Terms: conditions — Neuroendocrine Tumors; COVID-19; Coronavirus Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A huge number of initiatives about COVID-19 are ongoing and a growing number of publications regard the correlation between cancer patients in general and SARS-CoV-2 infection. Although it has been reported that cancer patients are at a higher risk of SARS-CoV-2 infection and COVID-19 complications, data collection about cases of NEN patients SARS-CoV-2 positive are scattered and related to single countries or institutions. Because of that and due to the rarity and heterogeneity of NEN it will be hard to have homogeneous, reliable, representative and reproducible data for drawing adequate clinical recommendations about NEN patients and COVID-19.

Therefore we propose a global collection of data through an international database to describe and monitor NEN patients with SARS-CoV-2 infection. This retrospective/prospective collection of data can create a solid basis to check frequence of events, clinical management, clinical outcome, demographic, geographical, clinical and biological correlations. This will be helpful for the clinical and scientific community to get reliable information for a homogeneous clinical management of NEN patients during COVID-19 pandemic.

The main goal is to get the as wide as possible representativity of the world situation.

DETAILED DESCRIPTION:
At the end of December 2019, several cases of pneumonia of unknown origin were diagnosed in Wuhan, in the province of Hubei, China. These cases have been linked to a new beta-coronavirus (COVID-19), identified with RT-PCR method from samples taken from the bronchoalveolar samples of a patient with pneumonia of unknown etiology in the Wuhan Jinyintan hospital. Severe acute respiratory coronavirus 2 syndrome (SARS-CoV-2) has spread rapidly worldwide causing a pandemic.

Cancer patients are considered at greater risk of viral infection and its complications, including SARS-CoV-2. Certain types of cancer, such as thoracic cancers, and underlying clinical conditions, for instance concomitant immunosuppressive therapies or immune-related comorbidities, are factors potentially predisposing to an increased risk of infection and eventually complications of COVID-19.

In this context, it is difficult to understand where and how to identify patients with neuroendocrine neoplasia (NEN).

We propose a global collection of data through an international database to describe and monitor NEN patients with COVID-19. This retrospective/prospective collection of data can create a large basis to check frequency of events, clinical management, clinical outcome, demographic, geographical, clinical and biological correlations.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 y.o.
* Patients with a NEN of any type with a positive SARS-CoV-2 swab (RT-PCR).
* Patients with SARS-CoV-2 positivity (RT-PCR) who are asymptomatic or with symptoms/signs of COVID-19.
* Patients with a NEN on active treatment.
* Patients with macroscopic evidence of NEN or with no evidence of NEN (if they received surgical +/- locoregional non-surgical treatments within the last 2 months)
* Able to provide signed written informed consent

Exclusion Criteria:

* Patients with NEN and symptoms suspected for COVID-19 who did not undergo SARS-CoV-2 swab (RT-PCR).
* Patients with small cell lung cancer.
* Patients with non-pure NEN (e.g. MiNEN).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a NEN of any type with a positive SARS-CoV-2 swab (RT-PCR).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-06-15 (Actual); Primary Completion 2023-12-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Correlation between clinical parameters and SARS-CoV-2 infection | 01/2020 - 12/2020
  To evaluate the correlation between SARS-CoV-2 infection and the following parameters: major comorbidities, severe overall events (including death), chemotherapy for neuroendocrine tumor (NET), chemotherapy for neuroendocrine carcinoma (NEC), everolimus therapy, immunotherapy, peptide receptor radionuclide therapy (PRRT) and surgery or radiotherapy within the last 2 months.
Clinical outcome of SARS-CoV-2 Infection | 01/2020 - 12/2020
  To evaluate the impact of SARS-CoV-2 Infection in NEN patients

SECONDARY OUTCOMES:
major demographic features | 01/2020 - 12/2020
  demographic features of SARS-CoV-2 infected NEN patients
type of NEN | 01/2020 - 12/2020
  Rate of grade, stage, status and primary site of NENs

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Fazio, M.D., Ph.D., Principal Investigator — European Institute of Oncology, IEO, IRCCS
Locations (1):
- European Institute of Oncology, IEO, IRCCS, Milan, MI, Italy

REFERENCES:
- [Background] Zhu N, Zhang D, Wang W, Li X, Yang B, Song J, Zhao X, Huang B, Shi W, Lu R, Niu P, Zhan F, Ma X, Wang D, Xu W, Wu G, Gao GF, Tan W; China Novel Coronavirus Investigating and Research Team. A Novel Coronavirus from Patients with Pneumonia in China, 2019. N Engl J Med. 2020 Feb 20;382(8):727-733. doi: 10.1056/NEJMoa2001017. Epub 2020 Jan 24. PMID 31978945
- [Background] Yu J, Ouyang W, Chua MLK, Xie C. SARS-CoV-2 Transmission in Patients With Cancer at a Tertiary Care Hospital in Wuhan, China. JAMA Oncol. 2020 Jul 1;6(7):1108-1110. doi: 10.1001/jamaoncol.2020.0980. PMID 32211820
- [Background] Al-Shamsi HO, Alhazzani W, Alhuraiji A, Coomes EA, Chemaly RF, Almuhanna M, Wolff RA, Ibrahim NK, Chua MLK, Hotte SJ, Meyers BM, Elfiki T, Curigliano G, Eng C, Grothey A, Xie C. A Practical Approach to the Management of Cancer Patients During the Novel Coronavirus Disease 2019 (COVID-19) Pandemic: An International Collaborative Group. Oncologist. 2020 Jun;25(6):e936-e945. doi: 10.1634/theoncologist.2020-0213. Epub 2020 Apr 27. PMID 32243668
- [Background] Liang W, Guan W, Chen R, Wang W, Li J, Xu K, Li C, Ai Q, Lu W, Liang H, Li S, He J. Cancer patients in SARS-CoV-2 infection: a nationwide analysis in China. Lancet Oncol. 2020 Mar;21(3):335-337. doi: 10.1016/S1470-2045(20)30096-6. Epub 2020 Feb 14. No abstract available. PMID 32066541

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan: version 1.0 (2020-05-11): https://cdn.clinicaltrials.gov/large-docs/01/NCT04444401/Prot_SAP_000.pdf
  • Study Protocol and Statistical Analysis Plan: version 1.1 (2020-06-09): https://cdn.clinicaltrials.gov/large-docs/01/NCT04444401/Prot_SAP_001.pdf
  • Informed Consent Form (2020-05-12): https://cdn.clinicaltrials.gov/large-docs/01/NCT04444401/ICF_002.pdf